CLINICAL TRIAL: NCT03501212
Title: Effect of Topical Anesthesia on Patient's Pain Discomfort and Radial Artery Spasm in Transradial Catheterization
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PMK-2018
Record Dates: First submitted 2018-03-21; First posted 2018-04-18 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Radial Artery Spasm
MeSH Terms: interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Active Comparator): EMLA group layer of 2.5 gr EMLA cream (standard adult dose) was applied to both wrists
  Interventions: Drug: Topical Anesthetic
- Placebo (Placebo Comparator): Placebo cream was applied to both wrists
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topical Anesthetic — EMLA Cream 2.5 gr applied to both wrists
  Arms: Interventional
Drug: Placebo — Placebo Cream 2.5gr applied to both wrist
  Arms: Placebo

SUMMARY:
This study evaluate topical anaesthesia application for 30 minutes before tranradial catheterization during cardiac catheterization can reduce pain and decrease radial artery spasm

DETAILED DESCRIPTION:
The incidence of Radial artery spasm (RAS) has varied from 5-30% RAS refers to friction between the artery and wires or guide catheters accompanied by a subjective feeling of pain.

EMLA anesthetic ointment (AO-Astra Zeneca) is an emulsion of lidocaine 2.5% and prilocaine 2.5% in a ratio of 1:1 by weight Previous study showed that EMLA cream can increase the success rate of femoral cannulation in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >18 years.
* Patients who was schedule to performed coronary angiogram

Exclusion Criteria:

Previous ipsilateral transradial approach Raynaud's syndrome ESRD History of sensitivity to local anesthetics Non-palpable redial pulse Abnormal Barbeau's test Local site infection Patient's refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-27 (Estimated); Primary Completion 2019-06-27 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Radial pain assessed during artery puncture | 30 min
  Record pain by visual analog score sub-scale 0(no pain)-10(max pain)

SECONDARY OUTCOMES:
Radial pain assessed 30 min after sheath removal | 4 hr post procedure
  Record pain by visual analog score
Number of puncture attempts | imediate post procedure
  Number of puncture attempts
Occurrence of radial artery spasm | during and post procedure up to 1 years
  NuNumber of radial artery spasm

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Bangkok, Thailand